CLINICAL TRIAL: NCT03633851
Title: Toric Intraocular Lens (IOL) Implantation Compared to Incisional Surgery to Correct Corneal Astigmatism as Part of Cataract Surgery - A Randomised Controlled Clinical Trial
Brief Title: Toric IOL vs Non-toric IOL With LRI for Corneal Astigmatism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ashford and St. Peter's Hospitals NHS Trust (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASPH2016-01
Record Dates: First submitted 2018-02-02; First posted 2018-08-16 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Corneal Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toric intraocular MX60T lens (Experimental): one eye will receive toric MX60T lens
  Interventions: Device: Toric intraocular MX60T lens
- Standard MX60 plus corneal incisions (Other): the other eye will receive standard MX60 lens with corneal incisions
  Interventions: Other: Standard MX60 plus corneal incisions

INTERVENTIONS:
Device: Toric intraocular MX60T lens — one eye will receive toric MX60T lens
  Arms: Toric intraocular MX60T lens
Other: Standard MX60 plus corneal incisions — the other eye will receive standard MX60 lens with corneal incisions
  Arms: Standard MX60 plus corneal incisions

SUMMARY:
The purpose of the study is to compare the astigmatism reducing effect of a toric intraocular lens (IOL) (model MX60T - Bausch & Lomb) with that of limbal relaxing incisional surgery combined with a non toric IOL (model MX60 - Bausch & Lomb) in patients with corneal astigmatism between 1.0 and 1.5 diopters and also the effect of cylinder reduction on patient's quality of vision.

DETAILED DESCRIPTION:
This is a randomised controlled trial with intra-patient comparison (bilateral study) in which study patients will be randomized by a medical statistician to the implantation of the toric intraocular lens (IOL) (model MX60T, Bausch & Lomb) in one eye and the non-toric IOL model MX60 plus LRI in the fellow eye.

During pre-operative examination, the patient will undergo:

* An ophthalmic examination including slit lamp biomicroscopy and retinal examination;
* Uncorrected and best-corrected visual acuity (UCVA and BCVA): monocular and binocular;
* Optical biometry with IOLMaster (Carl Zeiss Meditec);
* Orbscan corneal topography (Bausch and Lomb Orbscan IIz Corneal Analysis System);
* Quality of Vision (QoV) questionnaire score). It is a validated, Rasch-adjusted questionnaire in which patients are asked to rate 10 dysphotopsia items illustrated by standard photographs, scoring each item (0, 1, 2, 3) in relation to how frequent, severe, and bothersome their symptoms are (30 items in total).
* Catquest 9-SF cataract visual disability questionnaire. It is a Rasch-adjusted cataract visual disability questionnaire that asks patients to rate difficulty with a range of vision-related daily activities.

The appropriate cylinder power of the MX60T toric-IOL as well of its axis of implantation will be calculated with the calculator provided by the manufacturer Bausch + Lomb (https://trulign.toriccalculator.com).

Subsequently, the patient will undergo cataract surgery with IOL implantation under local anaesthesia.

The temporal self-sealing incision, injection of viscoelastic substance, capsulorhexis, phacoemulsification, irrigation/aspiration of cortical material and injection of viscoelastic substance into the capsular bag will be performed as standard procedure.

According to randomisation, each patient will receive the implantation of the MX60T toric-IOL in one eye and the MX60 non-toric IOL combined with limbal relaxing incisions (LRI) in the fellow eye.

The eye that will receive the toric-IOL will have the horizontal meridian marked preoperatively at the limbus in the sitting position with a blue marking pen and insulin syringe.

The IOL will be implanted via injector into the capsular bag using the manufacturers' recommended IOL loading and injection technique.

The toric-IOL will be rotated in the capsular bag so that the axis markers on the IOL will be aligned to the limbal markings (planned axis). Then, the viscoelastic substance will be aspirated thoroughly from the eye. Final refinement of axis position of the IOL will be undertaken after removal of viscoelastic material from the capsular bag to ensure that irrigation/aspiration of viscoelastic does not move the lens off axis.

The fellow eye will receive a temporal or an on-axis incision with limbal relaxing incision with a 600µm single-use steel blade combined with the MX60 non-toric IOL (http://www.lricalculator.com).

The interval between the first and second eye surgery will be recorded. The location and length of the LRIs will be made after calculation according to the Donnenfeld nomogram (www.lricalculator.com).

After one hour postoperatively, a photo of the toric-IOL in retroillumination will be taken to evaluate if IOL is on axis.

At six months and twelve months after the surgery performed in the second eye, patients will undergo assessement of:

* autorefraction;
* unaided and best-spectacle corrected visual acuity (monocular and binocular),
* optical biometry;
* corneal topography;
* photo of the toric-IOL in retroillumination (to evaluate if IOL is on axis);
* Catquest 9-SF cataract visual disability questionnaire;
* Quality of Vision (QoV) questionnaire score;
* Overall satisfaction with vision rating questionnaire (only at 6 months and 12 months). It will be obtained by asking patients to rate whether they were very satisfied, satisfied, neither satisfied nor unsatisfied, unsatisfied, or very unsatisfied.
* Dysphotopsia questionnaire. They are 4 questions regarding dysphotopsia symptoms: "Since your surgery, have you noticed any" halo, glare or dazzle, unwanted images, or shadows? Patients were asked to respond by indicating whether they had not experienced these symptoms at all ("none") or found them "barely noticeable," "annoying," or "debilitating."

Statistical analysis will be performed using SPSS for Macintosh software (version 20.0, International Business Machines Corp.). Normality distribution will be tested with the Shapiro-Wilk test; data will be considered normal if the p value is less than 0.05. The central tendency and statistical dispersion of each parameter will be recorded as the mean and standard deviation (SD) for normal data and as the median and interquartile difference for nonparametric data. The coordinates of keratometric cylinders and the centroids will be calculated according to the Alpins method. Double-angle polar plots will be used to display the astigmatism analysis (Excel 2011 for Macintosh, Microsoft Corp.).

The Student t test for paired samples and the Wilcoxon signed-rank test will be used for normal and nonparametric data, respectively, to compare the 2 related samples.

A statistically significant difference will be defined as a p value less than 0.05.

Any adverse event will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral cataract.
* Age 21 and older.
* Written informed consent to sequential bilateral surgery and participation in the study.
* Preoperative pupil size greater than or equal to 5.0 mm in the study eye.
* IOL power as predicted by biometry ranging from 6.0 D to 30.0 D in both eyes.
* Regular corneal astigmatism according to Orbscan topography.
* Postoperative corneal astigmatism between 0.90 D and 1.40 D in both eyes, as predicted by the Bausch + Lomb Toric Calculator (https://envista.toriccalculator.com).

Exclusion Criteria:

* Ocular comorbidity (corneal scars, amblyopia, retina, or optic nerve disease) that may reduce postoperative CDVA
* Reduced zonular or capsular stability (e.g. Marfan syndrome, previous eye trauma)
* Irregular corneal astigmatism on Orbscan topography

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-10-03 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Astigmatism reduction effect of toric intraocular lens (IOL) versus non-toric IOL with limbal relaxing incisions. | 6 months and 12 months
  Astigmatism reduction will be evaluated with optical biometry, corneal topography
Astigmatism reduction effect of toric intraocular lens (IOL) versus non-toric IOL | 6 months and 12 months
  Astigmatism reduction will be evaluated with manifest refraction, autorefraction

SECONDARY OUTCOMES:
Unaided visual acuity after toric intraocular lens (IOL) versus non-toric IOL with limbal relaxing incisions. | 6 months and 12 months
  Measurement of uncorrected visual acuity, monocular and binocular, will be done using a back-lit EDTRS chart placed at 4m. Although these assessments appear to have different units of measurements, but all the measurements will be in the same units of measure.
Best-spectacle corrected visual acuity after toric intraocular lens (IOL) versus non-toric IOL with limbal relaxing incisions. | 6 months and 12 months
  Measurement of best-spectacle corrected visual acuity, monocular and binocular, will be done using a back-lit EDTRS chart placed at 4m.
Quality of Vision | 6 months and 12 months
  Quality of Vision will be evaluated with the QoV (Quality of Vision) questionnaire score. It is a validated, Rasch-adjusted questionnaire in which patients are asked to rate 10 dysphotopsia items illustrated by standard photographs, scoring each item (0, 1, 2, 3) in relation to how frequent, severe, and bothersome their symptoms are (30 items in total).
Visual disability | 6 months and 12 months
  Visual disability will be evaluated with the Catquest 9-SF cataract visual disability questionnaire. It is a Rasch-adjusted cataract visual disability questionnaire that asks patients to rate difficulty with a range of vision-related daily activities.
Overall satisfaction | 6 months and 12 months
  Overall satisfaction will be evaluated with vision rating questionnaire. It will be obtained by asking patients to rate whether they were very satisfied, satisfied, neither satisfied nor unsatisfied, unsatisfied, or very unsatisfied.
Dysphotopsia | 6 months and 12 months
  Dysphotopsia will be evaluated with the Dysphotopsia questionnaire. They are 4 questions regarding dysphotopsia symptoms: "Since your surgery, have you noticed any" halo, glare or dazzle, unwanted images, or shadows? Patients were asked to respond by indicating whether they had not experienced these symptoms at all ("none") or found them "barely noticeable," "annoying," or "debilitating."

CONTACTS AND LOCATIONS:
Overall Officials: Vinod Gangwani, MBBS FRCS, Principal Investigator — Ashford and St. Peter's Hospitals NHS Trust
Locations (1):
- Dr Isaac John, Chertsey, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided